CLINICAL TRIAL: NCT01521026
Title: Cognitive Training for Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Elizabeth Twamley, Associate Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NARSAD Young Investigator
Record Dates: First submitted 2012-01-22; First posted 2012-01-30 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Other Primary Psychotic Disorders
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Training (Experimental): Cognitive training group
  Interventions: Behavioral: Cognitive Training
- Standard Pharmacotherapy (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Training — 12-week compensatory cognitive training in group format
  Arms: Cognitive Training

SUMMARY:
This research on cognitive training addresses the following questions:

1. Does cognitive training lead to improved cognition, functional abilities, psychiatric symptoms, treatment adherence, or quality of life in patients with psychoses?
2. What are the neurocognitive and non-cognitive factors that predict good outcomes following cognitive rehabilitation? In addition to verbal learning and memory, immediate verbal memory, vigilance, and executive functioning, the cognitive training intervention attempted to improve prospective memory ability (i.e., the ability to remember to do things in the future, such as take medications or attend a doctor's appointment).

ELIGIBILITY:
Inclusion Criteria:

* Primary psychotic disorder (including schizophrenia, schizoaffective disorder, psychotic mood disorder, or psychosis NOS)
* Age 18 or older
* Fluency in English

Exclusion Criteria:

* Dementia
* Neurological conditions affecting cognition
* Mental retardation
* Substance use disorder within the past month
* Participation in other intervention trials

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2003-09; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth W Twamley, PhD, Principal Investigator — UCSD
Locations (1):
- UCSD Outpatient Psychiatric Services, San Diego, California, United States

REFERENCES:
- [Derived] Twamley EW, Vella L, Burton CZ, Heaton RK, Jeste DV. Compensatory cognitive training for psychosis: effects in a randomized controlled trial. J Clin Psychiatry. 2012 Sep;73(9):1212-9. doi: 10.4088/JCP.12m07686. Epub 2012 Aug 7. PMID 22939029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants included 89 community-dwelling outpatients. Inclusion criteria were: primary psychotic disorder, age 18 or older, and fluency in English. Exclusion criteria were: dementia, neurological conditions affecting cognition, mental retardation, substance use disorder within the past month, and participation in other intervention trials.
Pre-assignment Details: Baseline data were collected before randomization.
Groups:
- Standard Pharmacotherapy: Standard pharmacotherapy with regular clinician
Period: Overall Study
Arm/Group | Cognitive Training | Standard Pharmacotherapy
Started | 38 | 31
Completed | 23 | 28
Not Completed | 15 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitive Training | Standard Pharmacotherapy | Total
Number analyzed (Participants) | 38 | 31 | 69
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 37 | 31 | 68
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (10.1) | 48.8 (8.7) | 46.3 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 | 24
  Male | 24 | 21 | 45
Region of Enrollment [Number; unit: participants]
  United States | 38 | 31 | 69

OUTCOME MEASURES:

1. Primary Outcome: UCSD Performance-based Skills Assessment Total Score (Measures Functional Capacity)
Description: Performance-based measure of functional capacity in five domains: Communication, Finance, Recreation Planning, Transportation, and Household Chores Scale ranges from 0-100. Subscales are summed to yield the total score. Higher scores represent better performance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard Pharmacotherapy: Standard pharmacotherapy with the regular clinician
Arm/Group | Cognitive Training | Standard Pharmacotherapy
Number analyzed (Participants) | 19 | 23
units on a scale | 82.7 (8.7) | 84.4 (8.0)

2. Secondary Outcome: Hopkins Verbal Learning Test Percent Retained
Description: Verbal list learning task with three learning trials and a delay trial. Percent retained refers to the percentage of items recalled at the delay trial, compared to the third learning trial.
  Score ranges from 0-100. Higher scores represent better performance.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cognitive Training | Standard Pharmacotherapy
Number analyzed (Participants) | 20 | 24
units on a scale | 93.4 (21.6) | 85.9 (19.4)

ADVERSE EVENTS:
Arm/Group | Cognitive Training | Standard Pharmacotherapy
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/31
Other Adverse Events (participants affected / at risk) | 0/38 | 0/31

LIMITATIONS AND CAVEATS:
* small sample size
* relatively short follow-up period
* significant dropout rate
* did not use an active control condition that matched CCT for therapist time or group involvement

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No